CLINICAL TRIAL: NCT00334906
Title: An Open-Label Exploratory Study With Memantine: Assessment of Selected Measures of Volumetric MRI and Cognition in Patients With Moderate Dementia of the Alzheimer's Type
Brief Title: Study of Memantine in Assessment of Selected Measures of Volumetric Magnetic Resonance Imaging (MRI) and Cognition in Moderate AD (Alzheimer's Disease)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEM-MD-15
Record Dates: First submitted 2006-06-06; First posted 2006-06-08 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2008-01

CONDITIONS: Alzheimer's Disease
Keywords: memantine; Alzheimer's disease; MRI; moderate Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

INTERVENTIONS:
Drug: memantine HCl

SUMMARY:
The purpose of this study is to characterize the progression of disease using volumetric MRI techniques and cognitive outcome measures in patients with moderate dementia of the Alzheimer's type treated with open-label memantine.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male or female patients at least 50 years of age (females at least 2 years postmenopausal)
* A diagnosis of probable AD [according to the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Associations (NINCDS-ADRDA) criteria] of moderate severity [Mini-Mental State Examination score between 15 and 20, inclusive]
* On a stable dose of Food and Drug Administration (FDA)-approved acetylcholinesterase inhibitor

Exclusion Criteria:

* Current Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (DSM-IV) Axis I disorder other than AD
* Previous imaging results not consistent with the diagnosis of AD
* Modified Hachinski Ischemia Score greater than 4
* Evidence of other neurologic disorders
* Inability to participate in MRI testing
* No clinically significant systemic disease
* A known or suspected history of alcohol or drug abuse in the past 10 years
* Taking excluded medication
* Previous treatment with commercial memantine

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2005-07; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Efficacy
Total brain atrophy on MRI

SECONDARY OUTCOMES:
Other measures of brain atrophy on MRI, change from baseline in selected cognitive measures assessing multiple cognitive domains including memory, attention, motor-speed, auditory comprehension, and verbal fluency
Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Forest Laboratories, Jersey City, New Jersey, United States